CLINICAL TRIAL: NCT01493336
Title: A Randomized, Open-label, Single Dose, Two-way Cross-Over Study to Investigate the Relative Bioavailability of Capecitabine in Rapid Disintegrating Tablets (RDT) Versus the Commercial Xeloda® Tablets Following Oral Administrations in Adult Patients With Solid Tumours
Brief Title: A Study of Capecitabine Rapid Disintegrating Tablets (RDT) Versus Commercial Xeloda in Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BP27931; 2011-005185-37 (EudraCT Number)
Record Dates: First submitted 2011-12-14; First posted 2011-12-15 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Breast Cancer, Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms | interventions — Capecitabine

ARMS (2):
- Capecitabine RTD (Experimental)
  Interventions: Drug: capecitabine RTD; Drug: capecitabine [Xeloda]
- Xeloda (Active Comparator)
  Interventions: Drug: capecitabine [Xeloda]

INTERVENTIONS:
Drug: capecitabine RTD — single oral dose
  Arms: Capecitabine RTD
Drug: capecitabine [Xeloda] — single oral dose
  Arms: Xeloda
Drug: capecitabine [Xeloda] — standard treatment

SUMMARY:
This randomized, open-label, two-way crossover study will evaluate the relative bioavailabilty and safety of capecitabine rapid disintegrating tablets (RDT) versus commercial Xeloda tablets in patients with colorectal or breast cancer. Patients will be randomized to a sequence of single oral doses of capecitabine RDT or Xeloda on Days 1 and 2 of a 14-day treatment cycle with Xeloda. Follow-up will be 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients,>/= 18 years of age
* Histological/cytological confirmation of colorectal or breast cancer
* Patient is ambulatory and has a Karnofsky performance status of > 70%
* Body surface area between 1.5 and 2.0 m2
* Either:
* Due to receive Xeloda as monotherapy or as combination therapy as per their treating physician's treatment plan, or
* Currently receiving Xeloda monotherapy and in the investigator's opinion able to tolerate study drug dose on Day 1 and Day 2

Exclusion Criteria:

* Any contraindication to Xeloda
* Received Xeloda in the 6 days prior to Day 1
* Subjects with organ allografts (other than autologous bone marrow transplant after high dose chemotherapy)
* Renal impairment
* Pregnant or lactating females
* Participation in an investigational drug study within 28 days prior to screening
* Lack of physical integrity of the upper gastrointestinal tract, or clinically significant malabsorption syndrome
* Serious uncontrolled intercurrent infections
* History of clinically significant coronary artery disease
* Concomitant treatment with warfarin
* Known dihydropyrimidine dehydrogenase deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2012-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Relative bioavailability: Area under the concentration-time curve (AUC) | Multiple sampling pre-dose to 6 hours post-dose

SECONDARY OUTCOMES:
Safety: Incidence of adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- Australia (2):
  - Adelaide, South Australia
  - Nedlands, Western Australia
- New Zealand (2):
  - Christchurch
  - Grafton
- United Kingdom (4):
  - Glasgow
  - Leeds
  - London
  - Newcastle upon Tyne